CLINICAL TRIAL: NCT06308354
Title: Colorectal Cancer Dataset in Xijing Hospital From 2011
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CRC dataset
Record Dates: First submitted 2024-02-18; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-01

CONDITIONS: Prognostic Cancer Model; Chemotherapy; Nutrition Related Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal cancer: Colorectal cancer patients are enrolled when patients were underwent surgeries.

SUMMARY:
To compare the differences of clinical pathological, treatment and prognosis in the guided subgroups in colorectal cancer, the investigator enrolled all the colorectal cancer patients who underwent surgery and were hospitalized in the Xijing hospital.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically confirmed colorectal adenocarcinoma, including hereditary colorectal cancer syndrome, such as Lynch syndrome and familial adenocarcinoma tumor polyposis, Peutz Jeghers syndrome, juvenile polyposis syndrome, and serrated polyposis syndrome;
* 2. Visit our center with complete medical records and pathological information;
* 3. Colorectal cancer patients diagnosed between 2013 and 2023.

Exclusion Criteria:

* 1. The patient has other colorectal malignancies other than adenocarcinoma;
* 2. Malignant tumors adjacent to organs invading the colon and rectum;
* 3. Malignant tumors from distant organs metastasize to the colon and rectum;
* 4. Benign colorectal lesions; 5. Patients with recurrent colorectal cancer.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients mainly comes from the western areas of China, and would accept the surgical procedures. Participate would be followed up every 6 months after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2048-01-01 (Estimated); Study Completion 2048-01-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | from date of diagnosis until the date of death from any cause, assessed up to 120 months
  to dead or lost to follow
DFS | from date of diagnosis until the first documented progression or recurrence, assessed up to 120 months
  disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
The investigators aim to explore the clinical characteristics of colorectal cancer patients in the Xijing hospital.

REFERENCES:
- [Derived] Cao S, Qiao Y, Wu L, Chen Q, Tian K, Li J, Xing C. Postoperative adjuvant chemotherapy in patients with stage II early onset colorectal cancer: exploration and discovery using real-world data and the SEER database. Front Oncol. 2025 May 30;15:1566569. doi: 10.3389/fonc.2025.1566569. eCollection 2025. PMID 40519292